CLINICAL TRIAL: NCT06970587
Title: Percutaneous Versus Transurethral Cystolithotripsy For The Management Of Bladder Calculi In The Pre-school Boys: Prospective Randomized Study
Brief Title: Percutaneous Versus Transurethral Cystolithotripsy For The Management Of Bladder Calculi In The Pre-school Boys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Hasan, Assistant Professor at Urology Department, Faculty of Medicine, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cystolithotripsy
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2019-02

CONDITIONS: Bladder Stone
MeSH Terms: conditions — Urinary Bladder Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): About 75 children suffering from bladder stone with a single bladder calculus ≤ 20 mm and managed by percutaneous cystolithotripsy (PCCL)
  Interventions: Procedure: percutaneous cystolithotripsy
- Group B (Active Comparator): About 75 children suffering from bladder stone with a single bladder calculus ≤ 20 mm and managed by transurethral cystolithotripsy (TUCL)
  Interventions: Procedure: percutaneous cystolithotripsy

INTERVENTIONS:
Procedure: percutaneous cystolithotripsy — to compare percutaneous cystolithotripsy with transurethral cystolithotripsy as minimally invasive surgical treatments for urinary bladder stones in pre-school age boys, and to assess the safety and the possible complications of both procedures
  Other Names: transurethral cystolithotripsy

SUMMARY:
Bladder stones are an uncommon condition in children, accounting for only 5% of urolithiasis in developed countries, whereas in developing nations, a greater number of children are affected due to the high incidence of urinary tract infections and inadequate nutrition, primarily a diet lacking in protein and rich in carbohydrates

DETAILED DESCRIPTION:
Bladder stones are typically categorized as either primary or secondary. Primary vesical stones are those not linked with urinary tract disease, and are typically found in children who experience episodes of diarrhea, as well as metabolic disorders resulting from inadequate hydration and nutrition.

Secondary bladder stones are linked to various urinary tract issues, such as obstruction at the bladder outlet, persistent infections, the presence of foreign objects, bladder diverticula, and neurological bladder problems.

The incidence of bladder stones is ten times more common in male than in female children, with children aged 1-5 years being more frequently affected, and the peak incidence occurs at 3 years of age.

The traditional treatment for bladder stones in children typically involves open cystolithotomy. The traditional open surgery has several inherent drawbacks, including a lengthy hospital stay, an unsightly suprapubic scar, the need for prolonged catheterization, the necessity for analgesic treatment, and the risk of post-operative wound infection .

Several minimally invasive treatment methods have been outlined, including transurethral cystolithotripsy (TUCL) and percutaneous cystolithotripsy (PCCL), with open cystolithotomy typically reserved for larger stones. In infants and toddlers, transurethral management bypasses abdominal invasion and its associated risks, such as paralytic ileus and fluid leakage.

However, this approach has limitations owing to the narrower urethral diameter compared to the larger diameter of the endoscopic equipment. In the past, percutaneous cystolithotripsy was commonly performed, but it was performed using larger equipment and has been replaced with transurethral cystolithotripsy. The use of mini-perc technology and smaller instruments for percutaneous stone removal is now competing with the transurethral procedure owing to recent advancements and reductions in percutaneous techniques and instruments.

The European guidelines for pediatric urology recommend endoscopy as an initial option for the management of bladder stones in children, with no distinction made between transurethral and percutaneous access methods. Undefined criteria indicate a lack of conclusive evidence to support one approach over the other, the reason for this is the insufficient number of prospective randomized trials which included a large number of patients comparing these techniques especially in this specific age group.

ELIGIBILITY:
Inclusion Criteria:

- All male preschool-aged patients (ages 1 to 6 years) who had a single bladder calculus measuring ≤ 20 mm in its longest dimensions diagnosed by ultrasonography or KUB.

Exclusion Criteria:

* Patients with proven bladder dysfunction, such as neurogenic bladder, bladder outlet obstruction, upper urinary tract stones requiring simultaneous ureteroscopy or percutaneous nephrolithotripsy,
* previous suprapubic procedure,
* severe skeletal malformation that prevents lithotomy position,
* bleeding tendency,
* active urinary tract infection

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Cystolithotripsy treatment | 45 minutes after the procedure begin
  Assessment of the Urinary Bladder condition of the patients after the Cystolithotripsy either successes or complications

SECONDARY OUTCOMES:
operative time | 45 minutes after the procedure begin
  Assessment of the time consumed of the Cystolithotripsy
Hospital stay duration | 24 hours after the Cystolithotripsy operation
  Assessment of the time required to stay in the hospital after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mahmoud Hasan, Assist.Prof., Principal Investigator — Urology Department,Faculty of Medicine,South Valley University,Qena,Egypt
Locations (1):
- South Valley University Hospitals, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Undecided